CLINICAL TRIAL: NCT03948672
Title: CleanHands Sensor Based System to Improve Hand Hygiene and Reduce Infection Trial
Brief Title: CleanHands Sensor Based System to Improve Hand Hygiene and Reduce Infection
Acronym: SHHRI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Microsensor Labs LLC (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); University of Louisville (Other); University of Chicago (Other); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 19.001; 4R44AG060848-02 (NIH)
Record Dates: First submitted 2019-05-10; First posted 2019-05-14 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Hand Hygiene; Infection
Keywords: hand hygiene; infection; sensor
MeSH Terms: conditions — Infections

STUDY DESIGN:
Intervention Model Description: Randomized, single blinded, crossover clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control-then-Intervention (Active Comparator): In each intensive care unit assigned to the Control-then-Intervention arm, all participants who regularly access the ICUs will wear the wristband while at work for 5 months. The functionality of the wristband will not be disclosed to the healthcare providers. Handwashing compliance data will be automatically collected, but data will not be shared with the healthcare providers or hospital management teams. After 5 months, a washout period of 2 months will be introduced to eliminate potential influences on healthcare providers' behaviors from the sensor system. Then, all healthcare providers will be educated on the functionalities of the CleanHands system with real time reminders now turned on. Healthcare providers will then have access to their own and unit-specific handwashing data. The unit manager and hospital administrators will be able to access all of these data and advanced analysis to make management decisions on infection reduction. This phase will last for 5 months.
  Interventions: Device: CleanHands System
- Intervention-then-Control (Active Comparator): In each intensive care unit assigned to the Intervention-then-Control arm, all participants who regularly access to the ICUs will be educated on the functionalities of the CleanHands system with real time reminders turned on. Healthcare providers will then have access to their own and unit-specific handwashing data. The unit manager and hospital administrators will be able to access all of these data and advanced analysis to make management decisions on infection control. This phase will last for 5 months. After 5 months, a washout period of 2 months will be introduced to eliminate potential influences on healthcare providers' behaviors from sensor system installation and implementation. Then, the real-time reminder functionality of the wristband will be turned off and no more education will be provided. Handwashing compliance data will be automatically collected but will not be shared with the healthcare providers. This process will last for 5 months.
  Interventions: Device: CleanHands System

INTERVENTIONS:
Device: CleanHands System — All participants who regularly access the ICUs will wear the CleanHands system wristband while at work for 5 months and the reminding functionality is turned on.

SUMMARY:
The purpose of this study is to determine if use of the CleanHands system can improve hand hygiene/personal protective equipment (PPE) compliance and reduce infections in the hospital ICUs through reminders to wash hands and use PPE as appropriate.

DETAILED DESCRIPTION:
Experimental design: The investigators plan to perform a randomized cross-over study at University of Louisville Hospital (ULH) ICUs from July 2019 to June 2020. The study will be submitted to the University of Louisville IRB for approval before any study activities are started.

Performance Site: University of Louisville Hospital. The ICU departments will be randomized to participate in either one of the two research arms: control-then-intervention arm or intervention-then-control arm.

Participants: All nurses, attending physicians, resident physicians, housecleaning staff, medical assistants, respiratory therapists, laboratory personnel (lab drawing) within experiment units.

Control-then-Intervention arm: In each intensive care unit assigned to the Control-then-Intervention arm, all participants who regularly access the ICUs will wear the wristband while at work for 5 months. The functionality of the wristband will not be disclosed to the healthcare providers. Handwashing compliance data will be automatically collected, but data will not be shared with the healthcare providers or hospital management teams. After 5 months, a washout period of 2 months will be introduced to eliminate potential influences on healthcare providers' behaviors from the sensor system. Then, all healthcare providers will be educated on the functionalities of the CleanHands system with real time reminders now turned on. Healthcare providers will then have access to their own and unit-specific handwashing data. The unit manager and hospital administrators will be able to access all of these data and advanced analysis to make management decisions on infection reduction. This phase will last for 5 months. All personnel will be educated not to discuss the functionalities of CleanHands system with their co-workers to ensure adequate blinding.

Intervention-then-Control arm: In each intensive care unit assigned to the Intervention-then-Control arm, all participants who regularly access to the ICUs will be educated on the functionalities of the CleanHands system with real time reminders turned on. Healthcare providers will then have access to their own and unit-specific handwashing data. The unit manager and hospital administrators will be able to access all of these data and advanced analysis to make management decisions on infection control. This phase will last for 5 months. After 5 months, a washout period of 2 months will be introduced to eliminate potential influences on healthcare providers' behaviors from sensor system installation and implementation. Then, the real-time reminder functionality of the wristband will be turned off and no more education will be provided. Handwashing compliance data will be automatically collected but will not be shared with the healthcare providers. The unit manager and hospital administrators will now be blinded to the handwashing compliance results. This process will last for 5 months.

Data collection: Handwashing compliance data are automatically collected by CleanHands. These data include all handwashing opportunities (defined as when a wristband is in pre-set proximity of the controller for 5 seconds or more), total cleaning solution dispensing counts, rates of

ELIGIBILITY:
Inclusion Criteria:

* All nurses, attending physicians, resident physicians, housecleaning staff, medical assistants, respiratory therapists, laboratory personnel (lab drawing) within experiment units.
* At least 18 years old
* Consent to participate in this study

Exclusion Criteria:

* Refusal to participate in this study
* Any reason that makes the participant not able to wear the CleanHands wristband

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-08-29 (Actual)

PRIMARY OUTCOMES:
hand hygiene compliance rate | 12 months
  percentage of qualified hand hygiene events divided by total hand hygiene opportunities.

SECONDARY OUTCOMES:
ICU infection rates | 12 months
  Catheter Associated Urinary Tract Infection (CAUTI), Central Line Associated Blood Stream Infection (CLABSI), C Diff, Bloodstream MRSA, Surgical Site Infection (SSI), Vancomycin Resistant Enterococcus (VRE), multiple drug resistant pseudomonas, Acinetobacter, Enterobacteriaceae, Carbapenem Resistant Enterobacteriaceae (CRE), and Carbapenem Resistant Organisms (CRO) rates.

CONTACTS AND LOCATIONS:
Overall Officials: Jiapeng Huang, MD, PhD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville Health, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.

REFERENCES:
- [Derived] Xu Q, Liu Y, Cepulis D, Jerde A, Sheppard RA, Reichle W, Scott L, Oppy L, Stevenson G, Bishop S, Clifford SP, Liu P, Kong M, Huang J. Hand hygiene behaviours monitored by an electronic system in the intensive care unit - a prospective observational study. J Hosp Infect. 2022 May;123:126-134. doi: 10.1016/j.jhin.2022.01.017. Epub 2022 Feb 2. PMID 35122887